CLINICAL TRIAL: NCT00662493
Title: The Effect of Specific Versus Generalised Quadriceps Exercise on Neural Control of the Vasti
Brief Title: A Comparison of Two Exercise Programs on Knee Motor Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Professor Kim Bennell, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 020077
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Knee Pain; Patellofemoral Pain
Keywords: knee pain; exercise; rehabilitation
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Motor control retraining program
  Interventions: Behavioral: Motor control retraining program; Behavioral: Quadriceps strengthening program

INTERVENTIONS:
Behavioral: Motor control retraining program — Specific retraining of VMO activation in a low-load situation,and progressed to integrate more functional positions. Use of dual channel biofeedback was incorporated
Behavioral: Quadriceps strengthening program — 4 exercises focused on quadriceps strengthening commencing at a resistance of 60% 1 repetition maximum. Each exercise was performed for 3 sets of 10 repetitions

SUMMARY:
Pain at the front of the knee is a common condition treated by physical therapists. Treatment may consist of generalised strengthening exercises directed at the quadriceps muscle or specific retraining aimed at restoring motor control at the knee. This study compared these two exercise programs in a group of people who were painfree at the time to evaluate their effect on motor control. It was hypothesised that only the motor retraining program would influence motor control at the knee.

ELIGIBILITY:
Inclusion Criteria:

* aged between 16-40 years, with the upper age limit to reduce the likelihood of osteoarthritic changes in the patellofemoral joint
* a self-reported history of anterior or retropatellar knee pain with insidious onset of symptoms and with at least one episode of pain in the past 12 months where pain was aggravated by at least two of the following: prolonged sitting, stairs, squat, running, kneeling and hopping/jumping
* currently asymptomatic for at least 8 weeks prior to assessment
* delay in the onset of VMO EMG relative to that of VL of greater than 10 ms during either the ascent or descent of a stair stepping task

Exclusion Criteria:

* current knee pain
* history of knee surgery or other knee injury in previous 12 months
* physiotherapy treatment for knee pain in the past 12 months
* history of patellar dislocation/subluxation
* clinical evidence of meniscal lesion, ligamentous instability, traction apophysitis around the patellofemoral complex, patellar tendon pathology, chondral damage, osteoarthritis and spinal referred pain
* current lower limb pathology affecting their ability to satisfactorily complete the testing or exercise protocol
* current use of non-steroidal anti-inflammatory or corticosteroid drugs
* inability to communicate and comprehend written or verbal instructions in English

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
latency between the onset of VMO electromyographic activity relative to that of VL during stair ascent and stair descent measured using surface electrodes | 6 weeks with 8 week followup

SECONDARY OUTCOMES:
Concentric and eccentric quadriceps muscle strength as assessed by isokinetic dynamometry | 6 weeks with 8 week followup

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Bennell, PhD, Principal Investigator — University of Melbourne; Kim Bennell, Principal Investigator — University of Melbourne; Kim Bennell, PhD, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Bennell K, Duncan M, Cowan S, McConnell J, Hodges P, Crossley K. Effects of vastus medialis oblique retraining versus general quadriceps strengthening on vasti onset. Med Sci Sports Exerc. 2010 May;42(5):856-64. doi: 10.1249/MSS.0b013e3181c12771. PMID 19997004